CLINICAL TRIAL: NCT01585636
Title: A Phase Ia, Randomized, Placebo-Controlled, Single-Dose, Double-Blind, Dose-Escalation Study to Evaluate Safety, Tolerability and Pharmacokinetics of SQ109 in Normal, Healthy Male and Female Volunteers
Brief Title: Escalating Single-dose Safety, Tolerability, and Pharmacokinetics of SQ109 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sequella, Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SQ109-CP001
Record Dates: First submitted 2012-04-20; First posted 2012-04-26 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Tuberculosis
Keywords: SQ109; Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- 5 mg dose group (Experimental): 8 subjects: 6 received active drug, 2 received matching placebo
  Interventions: Drug: SQ109
- 10 mg dose group (Experimental): 8 subjects: 6 received active drug, 2 received matching placebo
  Interventions: Drug: SQ109
- 20 mg dose group (Experimental): 8 subjects: 6 received active drug, 2 received matching placebo
  Interventions: Drug: SQ109
- 50 mg dose group (Experimental): 8 subjects: 6 received active drug, 2 received matching placebo
  Interventions: Drug: SQ109
- 100 mg dose group (Experimental): 8 subjects: 6 received active drug, 2 received matching placebo
  Interventions: Drug: SQ109
- 200 mg dose group (Experimental): 8 subjects: 6 received active drug, 2 received matching placebo
  Interventions: Drug: SQ109
- 300 mg dose group (Experimental): 8 subjects: 6 received active drug, 2 received matching placebo
  Interventions: Drug: SQ109
- Food effect group (Experimental): 6 Subjects received single, 300 mg SQ109 after high-fat, high-calorie meal.
  Interventions: Drug: SQ109

INTERVENTIONS:
Drug: SQ109 — Single oral dose

SUMMARY:
This is a phase 1, "first in man" study to evaluate single oral doses (5-300 mg) of SQ109, a new investigational drug being developed for treatment of tuberculosis. If single doses are safe and well tolerated, subsequent studies will evaluate multiple daily doses in healthy volunteers and patients with pulmonary tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18 to 55 years of age.
2. Subject must be a healthy male or female volunteer (i.e., hematology, coagulation,clinical chemistries and urinalysis tests must be within normal, allowable limits).

   Clinical laboratory tests must be performed within 21 days of receiving first dose of study drug.
3. Body weight must be ± 20% of the ideal for height and estimated frame based on the 1983 Metropolitan Life Insurance Company table.
4. Subject must give voluntary written informed consent before any study related procedure is performed.
5. Female subjects will be postmenopausal, surgically sterile, or agree to use two forms of contraception from screening through 30 days after the dose of study drug. All female subjects of childbearing potential must have a negative urine pregnancy test at screening.
6. Male subjects must agree to use an acceptable barrier method for birth control from screening through 30 days after the dose of study drug.

Exclusion Criteria:

1. A history of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
2. Subject has been on an abnormal diet during the 4 weeks preceding the study. Abnormal diet is defined as a diet in which the subject has a significant change in eating habits (e.g., liquid diet only) and an unbalanced diet (e.g., protein only, high fat, low carbohydrate, etc.).
3. Subject has donated blood within 30 days or plasma within 14 days of study dosing.
4. Subject has participated in any clinical trial within 30 days prior to study initiation; herein, 30 days are defined as 30 days from the last dosing in a clinical trial
5. Subject has used any over-the-counter (OTC) medication, including vitamins, within 7 days prior to the study.
6. Subject has used any prescription medication within 14 days prior to the study.
7. Subject has been treated with any known CYP450 enzyme altering drugs such as azoles, antifungals, barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to the study.
8. Subject has a positive blood screen for HIV, hepatitis B surface antigen (HBsAg), or hepatitis C antibody and/or a positive urine screen for alcohol or drugs of abuse.
9. Subject has smoked or used tobacco products within 2 months prior to or during the study.
10. Subject has an uncontrolled intercurrent illness (i.e., active infection).
11. Subject has had major surgery within 4 weeks of study entry.
12. Subject has another serious medical or psychiatric illness that could, in the Investigator's opinion, interfere with the completion of treatment according to this protocol.
13. Subjects who are color-blind.
14. Subjects with QTc interval prolongation (> 450 msec) or a history of QTc interval prolongation.
15. Subjects with a history of alcohol abuse, drug and/or food allergies.
16. Subjects who intend to consume grapefruit juice during the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2006-09; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Safety | daily examinations for 7 days after single dose drug administration
  Compared to baseline measurements:
  Change in Hb, Hct, WBC count / differential, platelet count Change in serum chemistry parameters Change in visual acuity Alteration in color perception Changes in cranial, sensory or motor nerve function, and mental status (as defined by the mini mental status examination) Prolongation in QTc interval, and rhythm changes by electrocardiogram

SECONDARY OUTCOMES:
Pharmacokinetics of SQ109 in fasted subjects and effect of high-fat, high calorie meal on pharmacokinetics | pK samples collected for 96 hours post dose administration
  maximum serum concentration (Cmax) Time to Cmax (Tmax) Area under the curve (AUC) Volume of Distribution (Vz/F) Oral clearance (CL/F)

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles Phaes 1 Clinical Study Unit, Lenexa, Kansas, United States